CLINICAL TRIAL: NCT01747564
Title: A Study to Evaluate Pharmacokinetics of Mirabegron After Single and Multiple Oral Administration to Healthy Non-elderly Male and Female Chinese Subjects
Brief Title: A Study to Evaluate Absorption, Distribution and Elimination of Mirabegron After Oral Administration to Non-elderly Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 178-CL-093
Record Dates: First submitted 2012-12-10; First posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Healthy Subjects; Plasma Concentration of Mirabegron
Keywords: Pharmacokinetics; Mirabegron; Phase 1; YM178
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mirabegron group (Experimental)
  Interventions: Drug: YM178 (mirabegron)

INTERVENTIONS:
Drug: YM178 (mirabegron) — oral
  Other Names: mirabegron

SUMMARY:
The purpose of this study is to evaluate safety and absorption, distribution and elimination of mirabegron after oral administration to Chinese subjects.

DETAILED DESCRIPTION:
This study is an open-label study. The subjects will receive single administration of mirabegron in a fasted condition. After the non-dosing period, subjects will receive mirabegron for 8 days.

ELIGIBILITY:
Inclusion Criteria:

* Body weight: (male) over 50.0kg and less than 80.0kg (female) over 40.0kg and less than 70.0kg
* Body Mass Index: over 17.6 and less than 26.4 kg/m
* Chinese subjects
* Healthy judged by investigator or sub-investigator

Exclusion Criteria:

* Received any investigational drugs within 120 days before the screening assessment
* Donated 400 mL of whole blood within 90 days, 200 mL of whole blood within 30 days, or blood components within 14 days before the screening assessment
* Received medication within 7 days before hospital admission
* A deviation from the assessment criteria of physical examinations or laboratory tests at screening or upon admission
* History of drug allergies
* With renal, hepatic, gastrointestinal, heart, cerebrovascular or respiratory diseases
* Received mirabegron beforehand
* Glaucoma patient

Ages: 20 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profile for ASP015K (in plasma): Cmax, AUClast, AUCinf and AUC0-24h | Day 1-5 and Day 10, 11, 14-21
  Maximum concentration (Cmax), Area under the curve (AUC) from time 0 extrapolated to infinity (AUCinf), AUC from time of dosing to last quantifiable concentration (AUClast ), and AUC from time 0 to 24hr (AUC0-24h)

SECONDARY OUTCOMES:
Safety assessed by the incidence of adverse events, vital signs, lab-test and 12-lead ECGs | Through day 25

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Kyushu, Japan